CLINICAL TRIAL: NCT02328092
Title: Therapeutic Effect of Sacral Root Stimulation on Nocturnal Enuresis
Brief Title: A Double-blind Randomized Clinical Trial on the Efficacy of Magnetic Sacral Roots Stimulation for the Treatment of NE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rSMS in nocturnal enuresis
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real group (Active Comparator): The real group received biphasic rSMS using a Magstim Super Rapid (Magstim, Whitland, UK) stimulator connected to a 120-mm outer diameter figure-of-8 air film cooling coil positioned in the midline over the sacral vertebrae (approximately 5 cm above the natal cleft, which approximates to the level of S2). Stimulation was delivered at 15 Hz at 50% of maximum stimulator output (10 seconds on and 30 seconds off) with a total of 1500 pulses and the hand of the coil upward. The stimulation was repeated for 10 sessions, 5 sessions per week and 2 days off.
  Interventions: Device: rSMS in treatment of Nocturnal Enuresis
- Sham Group (Sham Comparator): The control group received sham rSMS stimulation using the same coil, the same session frequency, in the same setting, but the coil was tilted 90.
  Interventions: Device: rSMS in treatment of Nocturnal Enuresis

INTERVENTIONS:
Device: rSMS in treatment of Nocturnal Enuresis — Real rSMS (15 Hz at 50% of maximum stimulator output (10 seconds on and 30 seconds off) with a total of 1500 pulses and the hand of the coil upword. The stimulation was repeated for 10 sessions, 5 sessions per week and 2 days off. Sham rSMS received stimulation using the same coil, the same session frequency, in the same setting, but the coil was tilted 90.

SUMMARY:
The purpose of this study is to assess the efficacy of daily sacral root magnetic stimulation for 10 sessions in patients with nocturnal enuresis.Eligible patients were randomized to receive either real or sham repetitive sacral root magnetic stimulation (rSMS; 15 Hz with a total of 1500 pulses/session) for 10 sessions. Evaluation was performed before starting treatment, immediately after the 5th and 10th treatment session, and 1 month later, using frequency of enuresis/week, visual analogue scale (VAS) and Quality of life. Cortical excitability of upper and lower limbs were done before and after the end of sessions.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of daily sacral root magnetic stimulation for 10 sessions in patients with nocturnal enuresis. Eligible patients were randomized to receive either real or sham repetitive sacral root magnetic stimulation (rSMS; 15 Hz with a total of 1500 pulses/session) for 10 sessions. Evaluation was performed before starting treatment, immediately after the 5th and 10th treatment session, and 1 month later, using frequency of enuresis/week, visual analogue scale (VAS) and Quality of life. Cortical excitability of upper and lower limbs were done before and after the end of sessions.

ELIGIBILITY:
Inclusion Criteria:

* All subjects diagnosed as patients with primary monosymptomatic nocturnal enuresis according to the Diagnostic and statistical manual of mental disorders, 4th revised edn (DSM-IV)

Exclusion Criteria:

* We exclude any patient with pacemakers or any metallic devices
* Patients with evidence of urinary tract infection.

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the number of bedwetting/week | 2.5 months
  Measurment of number of bedwetting/week one month before session, session, after first and second week of stimulation and one month later

SECONDARY OUTCOMES:
Quality of life assessment | 1.5 month
  Assessment of Quality of life
VAS | 1.5 month
  Measurment of VAS

REFERENCES:
- [Derived] Khedr EM, Elbeh KA, Abdel Baky A, Abo-Elfetoh N, El-Hammady DH, Korashy F. A double-blind randomized clinical trial on the efficacy of magnetic sacral root stimulation for the treatment of Monosymptomatic Nocturnal Enuresis. Restor Neurol Neurosci. 2015;33(4):435-45. doi: 10.3233/RNN-150507. PMID 26409403